CLINICAL TRIAL: NCT01011335
Title: A Randomized, Multi-Center Trial to Evaluate the Safety & Immunogenicity of Staphylococcus Aureus Toxoids, rAT and rLukS-PV, in Healthy Volunteers
Brief Title: Staphylococcus Aureus Toxoids Phase 1-2 Vaccine Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Nabi Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IDCRP-035/Nabi-6801; Nabi-W81XWH-09-2-0151; USAMRAA Grant #DR081318P1
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Staphylococcus Aureus
Keywords: Staphylococcus aureus; Skin and soft tissue infection; Methicillin-resistant Staphylococcus aureus; Recombinant alpha-toxoid (rAT); Recombinant LukS subunit of Panton-Valentine Leukocidin (rLukS-PV)
MeSH Terms: conditions — Staphylococcal Infections; Soft Tissue Infections | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Vaccine (Experimental): Monovalent rAT or Monovalent rLukS-PV or Bivalent rLukS-PV / rAT
  Interventions: Biological: Monovalent rAT; Biological: Monovalent rLukS-PV; Biological: Bivalent rLukS-PV / rAT
- Placebo with Alum (Placebo Comparator)
  Interventions: Biological: Placebo with adjuvant
- Saline Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Monovalent rAT — 10, 25, 50 or 100 μg
  Arms: Active Vaccine
Biological: Monovalent rLukS-PV — 10, 25, 50 or 100 μg
  Arms: Active Vaccine
Biological: Bivalent rLukS-PV / rAT — 10, 25 or 50 μg
  Arms: Active Vaccine
Biological: Placebo with adjuvant — Placebo with adjuvant
  Arms: Placebo with Alum
Biological: Placebo — Placebo saline
  Arms: Saline Placebo

SUMMARY:
This study involves the use of investigational vaccines. A vaccine is a medicine that causes the body to make antibodies. Antibodies help destroy foreign substances that enter the body. The purpose of this study is to find the right dose of a new vaccine that is safe and produces a good immune response (how well your body recognizes and defends itself against harmful foreign substances). There are two Staphylococcus aureus toxoids (components or antigens) under investigation in this study; one of them is a protein known as rAT and the other is a protein known as rLukS-PV. They are being developed to see if they are effective at preventing infections caused by the bacteria Staphylococcus aureus.

DETAILED DESCRIPTION:
Staphylococcus aureus is a leading cause of skin and soft tissue infections. Antibiotic resistance, such as seen with new community-acquired methicillin-resistant strains, presents a major challenge in treating and preventing these infections. Therefore, a preventative vaccine is considered a potentially better approach.

This study assesses the safety and immunogenicity of monovalent and bivalent S. aureus vaccine components. Healthy adult subjects will be randomized to receive 1 dose of monovalent or bivalent toxoid vaccine, or placebo in a dose escalation schedule.

Antigen-specific antibody will be measured by ELISA in sera collected for three months after injection. Safety data will be collected as 7 day reactogenicity diaries after each injection, adverse events and Staphylococcus aureus and skin and soft tissue infections will be collected through Day 84, and serious adverse events and chronic illnesses will be collected for the full 6 month study period.

To evaluate the possible utility of booster doses, the cohort receiving the highest dose of bivalent antigen will have a 2nd dose administered at Day 84, with a new 7-day reactogenicity diary and sera collected after the 2nd dose. All subjects will be followed up with a 6 month phone call after vaccination or booster.

The total subject observation period will be for 24 weeks from Day 0, plus 12 additional weeks for the cohorts that receive a 2nd dose. With a recruitment period of 4 months, the study duration is expected to be approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females, DoD beneficiaries, including active duty members, 18-55 years of age.
* Negative urine pregnancy test for female subjects of child bearing potential (negative test within 24 hours prior to investigational product injection) or documented surgical sterility.
* Female subjects of child-bearing potential must use an acceptable method of birth control, as determined by the PI.
* Willingness to participate in this study as evidenced by written informed consent.

Exclusion Criteria:

* Prior receipt of S. aureus rAT or rLukS-PV
* Known S. aureus infection requiring medical treatment within the 3 months prior to investigational drug product injection
* Known active viral or bacterial infection
* Seropositivity for HIV infection
* Known or suspected abuse of prescribed or illicit drugs, or alcohol in the past year
* Use of any new medications (except oral contraceptives, over-the-counter medications, or vitamin supplements) within the 7 days prior to investigational drug product injection
* Use of investigational drugs, vaccines, or devices during the study or within the 30 days prior to each dose of investigational drug product injection, or anticipated use of such items during the study
* Use of systemic steroids (any dose) or high daily dose inhaled steroids within the last month. Use of low or medium daily dose inhaled, intranasal, or low potency topical steroid creams/ointments is allowed unless such medication was begun within the previous 7 days.
* History of a bleeding or coagulation disorder; or use of anti-coagulant medications within 7 days prior to investigational product injection
* Actively breastfeeding
* Presence of grade I or higher abnormality in laboratory or vital signs parameter at time of screening
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Landrum, MD, Principal Investigator — Infectious Disease Clinical Research Program, Uniformed Services University of the Health Sciences; Paul Kessler, MD, Principal Investigator — Nabi Biopharmaceuticals
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were recruited from two clinical sites: San Antonio Military Medical Center, San Antonio, TX and Naval Medical Center, Portsmouth, VA between August 2010 and February 2011.
Pre-assignment Details: Subjects who consented to the study but who were not randomized were those who either failed screening due to abnormal baseline laboratory results, or who met screening criteria but became ineligible to receive a study injection or were unavailable at the time of injection. Subjects who were unavailable at the time of injection were replaced.
Groups:
- Monovalent rAT 10 ug Dose: Intramuscular; Monovalent rAT : 10 μg; single timepoint
- Monovalent rAT 25 ug Dose: Intramuscular; Monovalent rAT : 25 μg; single timepoint
- Monovalent rAT 50 ug Dose: Intramuscular; Monovalent rAT : 50 μg; single timepoint
- Monovalent rAT 100 ug Dose: Intramuscular; Monovalent rAT : 100 μg; single timepoint
- Monovalent rLukS 10 ug Dose: Intramuscular; Monovalent rLukS-PV : 10 μg; single timepoint
- Monovalent rLukS 25 ug Dose: Intramuscular; Monovalent rLukS-PV : 25 μg; single timepoint
- Monovalent rLukS 50 ug Dose: Intramuscular; Monovalent rLukS-PV : 50 μg; single timepoint
- Monovalent rLukS 100 ug Dose: Intramuscular; Monovalent rLukS-PV : 100 μg; single timepoint
- Bivalent rAT/rLukS 10 ug Dose: Intramuscular; Bivalent rAT/rLukS : 10 μg; single timepoint
- Bivalent rAT/rLukS 25 ug Dose: Intramuscular; Bivalent rAT/rLukS : 25 μg; single timepoint
- Bivalent rAT/rLukS 50 ug Dose: Intramuscular; Bivalent rAT/rLukS : 50 μg; single timepoint
- Alum Placebo: Intramuscular; Alum placebo : 10, 25, 50, 100 μg; single timepoint
- Normal Saline Placebo: Intramuscular; Saline Placebo : 10, 25, 50, 100 μg; single timepoint
Period: Overall Study
Arm/Group | Monovalent rAT 10 ug Dose | Monovalent rAT 25 ug Dose | Monovalent rAT 50 ug Dose | Monovalent rAT 100 ug Dose | Monovalent rLukS 10 ug Dose | Monovalent rLukS 25 ug Dose | Monovalent rLukS 50 ug Dose | Monovalent rLukS 100 ug Dose | Bivalent rAT/rLukS 10 ug Dose | Bivalent rAT/rLukS 25 ug Dose | Bivalent rAT/rLukS 50 ug Dose | Alum Placebo | Normal Saline Placebo
Started | 11 | 12 | 12 | 12 | 13 | 12 | 12 | 12 | 12 | 12 | 12 | 22 | 22
Completed | 10 | 11 | 11 | 10 | 12 | 11 | 9 | 10 | 10 | 12 | 6 | 21 | 19
Not Completed | 1 | 1 | 1 | 2 | 1 | 1 | 3 | 2 | 2 | 0 | 6 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Moved/deployed or no booster | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Monovalent rAT Doses: Monovalent rAT : 10, 25, 50 or 100 μg
- Monovalent rLukS-PV Doses: Monovalent rLukS-PV : 10, 25, 50 or 100 μg
- Bivalent rAT/rLukS-PV Doses: Bivalent rLukS-PV / rAT : 10, 25 or 50 μg
- Placebo Doses: Saline placebo or alum placebo
- Total: Total of all reporting groups
Arm/Group | Monovalent rAT Doses | Monovalent rLukS-PV Doses | Bivalent rAT/rLukS-PV Doses | Placebo Doses | Total
Number analyzed (Participants) | 47 | 49 | 36 | 44 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.0) | 31.1 (8.6) | 32.0 (8.6) | 32.9 (10.2) | 32.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 15 | 16 | 60
  Male | 32 | 35 | 21 | 28 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 6 | 6 | 27
  Not Hispanic or Latino | 38 | 43 | 30 | 38 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39 | 36 | 28 | 29 | 132
  Black | 6 | 7 | 7 | 10 | 30
  All Other | 2 | 6 | 1 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Safety Through Clinical Examinations, Clinical Laboratory Results, Self-reported Diary Reactogenicity Data and Adverse Event Reports
Description: Adverse events, local reactogenicity, and systemic reactogenicity were assessed through clinical examination by study providers, clinical lab results, as well as review of subject-completed diary
Time Frame: Up to 6 months
Measure: Number; unit: events
Groups:
- Monovalent rAT Doses: Monovalent rAT 10µg, 25µg, 50µg, 100µg
- Monovalent rLukS Doses: Monovalent rLukS 10µg, 25µg, 50µg, 100µg
- Bivalent rAT/rLukS Doses: rAT/rLukS 10µg, 25µg, 50µg
- Placebo Doses: Alum placebo and Saline placebo
Arm/Group | Monovalent rAT Doses | Monovalent rLukS Doses | Bivalent rAT/rLukS Doses | Placebo Doses
Number analyzed (Participants) | 47 | 49 | 36 | 44
events
  Adverse Events | 37 | 40 | 28 | 36
  Local or Systemic Reactogenicity Events | 31 | 41 | 29 | 24

2. Primary Outcome: Immunogenicity: Geometric Mean Concentrations After First Injection, Completer Population
Description: Immunogenicity is the ability of a particular substance, such as an antigen or epitope, to provoke an immune response in the body of a human or animal. Immunogenicity was determined on the basis of anti-rAT and anti-rLukS-PV IgG concentrations assessed by enzyme-linked immunosorbent assay (ELISA) in sera from blood samples collected on Days 0 (baseline), 14, 28 and 84 for those receiving a single dose of vaccine. For those receiving a second dose of vaccine, immunogenicity assessments were also conducted on Days 98 and 112. Immunogenicity was evaluated using the following metrics: geometric mean concentrations (GMCs), geometric mean fold increase (GMFIs) and seroresponse status. Seroresponse variables are normally defined in terms of exceeding a threshold.
Time Frame: Up to 3 months
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | rAT 10 µg | rAT 25 µg | rAT 50 µg | rAT 100 µg | rAT/rLukS 10 µg (for rAT) | rAT/rLukS 25 µg (for rAT) | rAT/rLukS 50 µg (for rAT) | Alum Placebo (for rAT) | Saline Placebo (for rAT) | rLukS 10 µg | rLukS 25 µg | rLukS 50 µg | rLukS 100 µg | rAT/rLukS 10 µg (for rLukS) | rAT/rLukS 25 µg (for rLukS) | rAT/rLukS 50 µg (for rLukS) | Alum Placebo (for rLukS) | Normal Saline Placebo (for rLukS)
Number analyzed (Participants) | 11 | 11 | 12 | 9 | 10 | 11 | 12 | 21 | 20 | 11 | 11 | 12 | 11 | 10 | 11 | 12 | 21 | 20
μg/mL
  Day 0 | 27.9 [18.7 to 41.7] | 20.7 [11.3 to 37.9] | 16.0 [9.4 to 27.3] | 25.4 [14.9 to 43.4] | 20.9 [12.0 to 36.5] | 32.3 [19.2 to 54.5] | 17.0 [11.7 to 24.8] | 18.5 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.36 | 20.9 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.17 | 12.1 [6.81 to 21.48] | 13.2 [6.68 to 26.06] | 13.1 [7.49 to 22.91] | 9.0 [4.33 to 18.74] | 10.4 [6.66 to 16.17] | 16.8 [8.19 to 34.23] | 17.7 [11.14 to 28.02] | 16.0 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.71 | 22.3 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.41
  Day 14 | 47.6 [29.4 to 77.0] | 157 [110.9 to 220.9] | 356 [173.8 to 731.1] | 261 [108.9 to 625.4] | 51.1 [27.9 to 93.7] | 116 [64.4 to 207.4] | 213 [141.2 to 320.3] | 20.9 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.46 | 20.5 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.27 | 35.7 [14.11 to 90.40] | 133 [63.16 to 278.5] | 91.7 [37.72 to 223.0] | 67.2 [27.82 to 162.4] | 29.0 [14.16 to 59.39] | 60.2 [22.53 to 161.1] | 108 [65.39 to 179.1] | 15.8 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.71 | 21.5 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.53
  Day 28 | 51.7 [30.9 to 86.4] | 185 [141.6 to 242.3] | 338 [172.8 to 659.4] | 232 [92.0 to 586.9] | 50.2 [28.4 to 88.8] | 129 [77.9 to 213.7] | 223 [145.2 to 342.8] | 19.4 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.43 | 19.5 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.32 | 39.8 [15.53 to 101.8] | 166 [78.57 to 352.6] | 103 [43.69 to 244.0] | 81.7 [34.20 to 195.1] | 31.2 [15.13 to 64.34] | 68.1 [27.19 to 170.5] | 108 [61.93 to 187.1] | 14.8 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.91 | 20.7 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.54
  Day 84 | 57.8 [34.5 to 96.9] | 159 [119.5 to 212.2] | 313 [176.9 to 553.5] | 223 [133.6 to 372.5] | 46.8 [26.4 to 82.8] | 111 [70.5 to 176.1] | 167 [96.9 to 289.2] | 18.8 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.46 | 19.6 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=2.13 | 39.6 [16.93 to 92.81] | 128 [61.02 to 267.1] | 85.0 [35.91 to 201.5] | 68.6 [29.02 to 162.0] | 29.4 [14.73 to 58.66] | 59.2 [25.66 to 136.6] | 82.5 [45.39 to 149.8] | 14.7 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.71 | 24.6 [NA to NA] — 95% confidence Intervals not available for this group due to insufficient number of participants with data. Standard deviations were calculated. SD=3.95
  Day 98 | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | 203 [NA to NA] — 95% confidence Intervals not available for this group at Day 98 due to insufficient number of participants with data. Standard deviations were calculated. SD=2.2 | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | 93.3 [NA to NA] — 95% confidence Intervals not available for this group at Day 98 due to insufficient number of participants with data. Standard deviations were calculated. SD=2.48 | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112.
  Day 112 | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | 116 [NA to NA] — 95% confidence Intervals not available for this group at Day 112 due to insufficient number of participants with data. Standard deviations were calculated. SD=6.27 | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | 57.6 [NA to NA] — 95% confidence Intervals not available for this group at Day 112 due to insufficient number of participants with data. Standard deviations were calculated. SD=6.09 | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112. | NA [NA to NA] — Arm did not receive booster and were not evaluated at Days 98 and 112.

ADVERSE EVENTS:
Arm/Group | Monovalent rAT 10µg Dose | Monovalent rAT 25µg Dose | Monovalent rAT 50µg Dose | Monovalent rAT 100µg Dose | Monovalent rLukS 10µg Dose | Monovalent rLukS 25µg Dose | Monovalent rLukS 50µg Dose | Monovalent rLukS 100µg Dose | Bivalent rAT/rLukS 10µg Dose | Bivalent rAT/rLukS 25µg Dose | Bivalent rAT/rLukS 50µg Dose | Alum Placebo | Normal Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12 | 0/12 | 0/13 | 0/12 | 1/12 | 0/12 | 0/12 | 1/12 | 2/12 | 0/22 | 1/22
Other Adverse Events (participants affected / at risk) | 7/11 | 10/12 | 10/12 | 9/12 | 9/13 | 12/12 | 9/12 | 10/12 | 7/12 | 8/12 | 12/12 | 19/22 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monovalent rAT 10µg Dose (N=11) | Monovalent rAT 25µg Dose (N=12) | Monovalent rAT 50µg Dose (N=12) | Monovalent rAT 100µg Dose (N=12) | Monovalent rLukS 10µg Dose (N=13) | Monovalent rLukS 25µg Dose (N=12) | Monovalent rLukS 50µg Dose (N=12) | Monovalent rLukS 100µg Dose (N=12) | Bivalent rAT/rLukS 10µg Dose (N=12) | Bivalent rAT/rLukS 25µg Dose (N=12) | Bivalent rAT/rLukS 50µg Dose (N=12) | Alum Placebo (N=22) | Normal Saline Placebo (N=22)
Alcoholism (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Astrocytoma Malignant (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac Chest Pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monovalent rAT 10µg Dose (N=11) | Monovalent rAT 25µg Dose (N=12) | Monovalent rAT 50µg Dose (N=12) | Monovalent rAT 100µg Dose (N=12) | Monovalent rLukS 10µg Dose (N=13) | Monovalent rLukS 25µg Dose (N=12) | Monovalent rLukS 50µg Dose (N=12) | Monovalent rLukS 100µg Dose (N=12) | Bivalent rAT/rLukS 10µg Dose (N=12) | Bivalent rAT/rLukS 25µg Dose (N=12) | Bivalent rAT/rLukS 50µg Dose (N=12) | Alum Placebo (N=22) | Normal Saline Placebo (N=22)
Haemoglobin decreased (Blood and lymphatic system disorders) | 3 | 1 | 7 | 9 | 1 | 1 | 3 | 3 | 3 | 2 | 2 | 3 | 6
Blood glucose increased (Blood and lymphatic system disorders) | 1 | 2 | 3 | 7 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 3 | 4
ALT increased (Blood and lymphatic system disorders) | 2 | 1 | 3 | 3 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 3 | 0
Blood glucose decreased (Blood and lymphatic system disorders) | 0 | 2 | 1 | 4 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Haemoglobin abnormal (Blood and lymphatic system disorders) | 1 | 0 | 1 | 3 | 0 | 2 | 4 | 0 | 1 | 0 | 0 | 2 | 1
AST increased (Blood and lymphatic system disorders) | 1 | 0 | 5 | 2 | 1 | 0 | 1 | 0 | 0 | 4 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 4 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2
Blood urea increased (Renal and urinary disorders) | 1 | 1 | 2 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Blood LDH increased (Blood and lymphatic system disorders) | 1 | 1 | 3 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1
WBC count increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 3
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Hypoglycaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Blood sodium increased (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Hyperglycaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Protein urine present (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
GERD (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Injection site swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Numbers in each of the dose arms were small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No